CLINICAL TRIAL: NCT04871087
Title: Narrow Band Green Light (NBGL) Effects on the Treatment of Anxiety During Psychotherapy Sessions: a Pilot Study
Brief Title: Green Light Effects on Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Green Light Study Center (Other)
Responsible Party: Principal Investigator, Paul Hart, Dr. Paul Hart, The Green Light Study Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 002
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: single arm assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allay lamp (narrow band green light) (Other): Comparing effects of NBGL vs. white light on anxiety level before and after psychotherapy treatment sessions.
  Interventions: Device: Green Light

INTERVENTIONS:
Device: Green Light — The Allay Lamp is a consumer product currently available and widely used in the US. It emits low intensity (1-10lux)narrow band (20nm) green light (peak wavelength 520nm) that is marketed as non-irritating to users. In that context, it is not a medical device and does not require a 510(k). However, we believe that light likely also has benefits for sleep. To better understand its effects,we are planning to conduct the proposed study. In that context, the Allay Lamp would be considered an investigational medical device because it has not been cleared or approved by FDA for the intended purpose of treating sleep. No FDA submission should be necessary for this study using 21 C.F.R. 812.3, because the Allay Lamp is a non-significant risk (NSR) device:
  It is not an implant It is not intended for use in supporting or sustaining human life The Allay Lamp provides a very low risk light-based therapy. The light provides no more risk than any other table lamp available on the market today.

SUMMARY:
The main goal of this study is to determine whether exposure to a narrow band of green light (NBGL) improves outcome of psychotherapy sessions for the treatment of anxiety.

This is a within-subject study design that examines NBGL effects (as compared to white light) on anxiety level and treatment success, as evaluated by the treating psychotherapist and the patient. For each participant, the study will consist of 8 therapy sessions, each lasting 60 minutes, in which light conditions will be presented in the following order

Session 1: White light, Session 2: white light, Session 3: NBGL (i.e., green light), Session 4: NBGL, Session 5: NBGL, Session 6: NBGL, Session 7: White light, Session 8: White light

Effects of lights (white vs.NBGL) on anxiety level will be evaluated at the beginning and end of each therapy session by the patient, using a validated questionnaire. At the end of each session, the treating psychotherapist will fill another evaluation form that summarizes her/his impression of the treatment success or lack of.

DETAILED DESCRIPTION:
Each patient is treated once a week and thus, study participation time is expected to last 8 weeks. Patients will self evaluate their anxiety level at the beginning and end of each of the 8 therapy sessions by completing the 20-questions State-Trait Anxiety Inventory (STAI Form Y-1).

Therapists will fill the following form after each of the 8 sessions:

Did you feel any difference while working with the patient in the green light as compared to regular room light?

Check all that apply:

* I was more focused
* I was more relaxed
* The patient was more relaxed
* The patient was more engaged
* The patient seemed more open
* The therapy progressed further

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anxiety
* Being a patient at the Delray Center
* Older than 18 and younger than 95
* Being able to communicate in English
* Willingness to sign informed consent

Exclusion Criteria:

* Co-morbid psychiatric conditions

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 1 year
  Changes in anxiety level, as measured by the STAI (State-Trait Anxiety Inventory)

CONTACTS AND LOCATIONS:
Locations (1):
- Delray Center for Healing, Delray Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided